CLINICAL TRIAL: NCT05343728
Title: The Role of Thromboelastographic Methods in Deciding Therapy on Moderate to Severe COVID-19
Brief Title: Thromboelastographic Methods in Deciding Therapy on Moderate to Severe COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andi Ade Wijaya Ramlan, Principal Investigator, Indonesia University
Other Study IDs: IndonesiaUAnes114
Record Dates: First submitted 2022-04-21; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: Thromboelastography; Blood coagulation disorder; Mortality; intensive care unit
MeSH Terms: conditions — COVID-19; Blood Coagulation Disorders | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thromboelastographic Methods: Patients whose coagulation profile were done by using a thromboelastography in addition to standard coagulation profile laboratory examination (thrombocyte count, PT, APTT, D-dimer, Fibrinogen)
  Interventions: Diagnostic Test: Thromboelastography; Diagnostic Test: Standard coagulation profile laboratory examination
- Standard coagulation profile laboratory examination: Patients whose coagulation profile were done by using a standard coagulation profile laboratory examination (thrombocyte count, PT, APTT, D-dimer, Fibrinogen)
  Interventions: Diagnostic Test: Standard coagulation profile laboratory examination

INTERVENTIONS:
Diagnostic Test: Thromboelastography — Thromboelastography was done by using TEG 5000 Hemostasis Analyzer (Haemonetics Corp., USA)
  Other Names: TEG 5000 Hemostasis Analyzer (Haemonetics Corp., USA)
  Groups: Thromboelastographic Methods
Diagnostic Test: Standard coagulation profile laboratory examination — Standard coagulation profile laboratory examination (platelets, PT/APTT, fibrinogen, and D-dimer) was performed by using Sysmex® CS-2500 and 5100 (Sysmex Corp., Japan)

SUMMARY:
This study is a prospective observational study that compares the anticoagulant therapy decision time among moderate and severe COVID-19 patients whose coagulation profiles were tested with thromboelastography (TEG) to those with a standard coagulation profile laboratory examination.

DETAILED DESCRIPTION:
A prospective observational study was conducted among moderate to severe COVID-19 patients in the High Care Unit and Intensive Care Unit at Kiara Ultimate, Cipto Mangunkusumo Hospital, Indonesia. We consecutively recruited 100 moderate and severe COVID-19 patients in the high and intensive care units.

Baseline characteristic data collection was carried out when the patient was admitted to the ICU or HCU. Venous blood was taken by nurses within 30 min of admission. The samples were sent to the centralized hospital laboratory for a standard hemostasis panel which consisted of platelets, PT/APTT, fibrinogen, and D-dimer. The hospital used Sysmex® CS-2500 and 5100 (Sysmex Corp., Japan) for coagulation tests by using plasma derived from centrifuged whole blood samples. Bedside TEG examination was done by using TEG 5000 Hemostasis Analyzer (Haemonetics Corp., USA) with 2.5 ml of a whole blood sample. Samples of patients with heparin thromboprophylaxis were given heparinase, which binds to heparin so that the coagulation profile can be assessed. Except for TEG, all patients received equal diagnostic tests and treatment, including anticoagulant therapy, as indicated according to the national guideline. A trained doctor from the research team recorded time from blood samples taken until the coagulation panel or TEG results were obtained. Test result timestamp, anticoagulation decision timestamp, mortality, and length of stay in higher care were objectively retrieved through online medical records.

We compared the result turnaround time, time to decision of anticoagulant therapy, and clinical outcomes (length of stay and 30-day mortality) between those who had TEG examination in addition to standard coagulation profile examination (thrombocyte count, PT, APTT, D-dimer, and fibrinogen) and those who had a standard coagulation profile laboratory examination only.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19 (Positive SARS-CoV-2 PCR test), 3. Moderate or severe symptoms (We defined moderate COVID-19 as patients with clinical signs of pneumonia with SpO2 >93% in room air and severe COVID-19 as pneumonia with SpO2 ≤93% in room air or ventilator support requirement), and 4. The family signed the informed consent

Exclusion Criteria:

1. History of blood clotting disorders (eg, hemophilia and Von Willebrand's disease),
2. Have contraindications to the administration of anticoagulants, for example:

   1. Platelet count < 25,000
   2. Has bleeding manifestations
   3. History of heparin allergy or heparin-induced thrombocytopenia
3. Pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was patients who had confirmed COVID-19 and underwent treatment at Cipto Mangunkusumo Hospital from October 2020 to March 2021. Subjects were eligible if they were adults (aged >18 years) who had positive SARS-CoV-2 nasopharyngeal swab examination with moderate to severe clinical symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Time to anticoagulant therapy decision | First day of admission in ICU/HCU
  Calculation of the time (minutes) required from blood sample was taken until the decision on anticoagulant therapy made by the supervisors

SECONDARY OUTCOMES:
Result turnaround time | First day of admission in ICU/HCU
  Calculation of the time (minutes) required from blood sample was taken until the examination result was done
Length of stay in higher care | During hospitalization
  Length of stay in intensive care unit and/or high care unit during admission
Mortality | 30 days after hospital admission
  Death within 30 days after admission to the intensive care unit and/or high care unit

CONTACTS AND LOCATIONS:
Overall Officials: Andi Ade Wijaya Ramlan, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided